CLINICAL TRIAL: NCT01977573
Title: A 24-week, Phase IIB, Randomized, Controlled, Parallel Group, Multi-center Study to Evaluate the Safety and Efficacy of GSK1278863 in Subjects With Anemia Associated With Chronic Kidney Diseases Who Are Not on Dialysis.
Brief Title: A Study to Evaluate Safety and Efficacy of GSK1278863 in Non-Dialysis Dependent (NDD) Subjects With Anemia Associated With Chronic Kidney Diseases (CKD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 113747
Record Dates: First submitted 2013-10-24; First posted 2013-11-06 (Estimated); Results first posted 2016-06-06 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-09

CONDITIONS: Anaemia
Keywords: Prolyl hydroxylase inhibitor; pharmacokinetics; GSK1278863; Anemia; hemoglobin; erythropoiesis stimulating agents; Chronic kidney disease
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — GSK1278863

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GSK1278863 (Experimental): Subjects will be administered GSK1278863 QD. Starting dose will be based on data from previous studies with GSK1278863 and dose-response modelling, as well as Baseline Hgb concentration. After 4 Week of fixed dose period, dose may be adjusted to achieve Hgb 9.0 to 10.5 g/dL
  Interventions: Drug: GSK1278863
- Control (Other): All subjects who are randomized to the Control arm will receive rhEPO (epoetins or their biosimilars, or darbepoetin) as necessary per standard of care, to maintain Hgb levels within the target range. The decision around whether a subject requires rhEPO, selection of the type of rhEPO and rhEPO dose should be based on Investigator clinical judgment, with the historical rhEPO dose (where applicable) and the current Hgb value being considered.
  Interventions: Drug: rhEPO

INTERVENTIONS:
Drug: GSK1278863 — Film-coated tablets containing 0.5 mg, 1 mg, 2 mg, 5mg or matching placebo
  Arms: GSK1278863
Drug: rhEPO — Locally sourced rhEPO. All subjects who are randomized to the Control arm will receive rhEPO (epoetins or their biosimilars, or darbepoetin) as necessary per standard of care, to maintain Hgb levels within the target range. The decision around whether a subject requires rhEPO, selection of the type of rhEPO and rhEPO dose should be based on Investigator clinical judgment, with the historical rhEPO dose (where applicable) and the current Hgb value being considered..
  Arms: Control

SUMMARY:
This study will be conducted in approximately 228 subjects with anemia associated with CKD who are not on dialysis. Two groups of subjects will be enrolled into the study: Group 1: recombinant human erythropoietin (rhEPO) naive subjects; Group 2: rhEPO users, who are currently receiving rhEPO. Subjects who are rhEPO naive will be randomized to receive either GSK1278863 once daily (QD) or rhEPO in a 3:1 fashion; subjects who are receiving an rhEPO before enrolling (rhEPO users) will be randomized in a 1:1 fashion to GSK1278863 QD or to the control arm. For those randomized to the control arm, the decision around whether the subject requires rhEPO, the selection of the type of rhEPO (if needed) and the choice of rhEPO dose to achieve and maintain Hgb concentrations within the target range should be based on Investigator clinical judgment, with the historical rhEPO dose and the current Hgb value being considered. The study consists of a screening phase of at least 4 weeks, a 24-week treatment phase and a follow-up visit that will occur approximately 4 weeks after completing treatment. It is anticipated that the data generated will enable selection of the starting dose(s) and optimize dose adjustment regimen(s) for Phase 3 clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Age: >=18 years of age. (Week -4 verification only)
* Gender: Female and male subjects. (Week -4 verification only) Females: If of childbearing potential, must agree to use one of the approved contraception methods, from Screening until completion of the Follow-up Visit OR Of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation, hysterectomy, or oophorectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea. Females on hormone replacement therapy (HRT) whose menopausal status is in doubt will be required to use one of the approved contraception methods if they wish to continue their HRT during the study. Otherwise they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.
* Corrected QT interval (QTc): Bazett's Correction of QT Interval (QTcB) <470 milliseconds (msec) or QTcB <480 msec in subjects with bundle branch block. There is no QTc criterion for subjects with a predominantly paced rhythm.
* CKD stage: Kidney Disease Outcomes Quality Initiative (KDOQI) CKD stages 3/4/5 defined by electronic estimated glomerular filtration rate (eGFR) using the CKD Epidemiology Collaboration (CKD-EPI) formula.
* Hgb: Group 1 (rhEPO naïve): Baseline Hgb of 8.0-11.0 g/dL (inclusive) (USA sites only: 8.0-10.0 g/dL, inclusive); Group 2 (rhEPO users): Baseline Hgb of 9.0-11.5 g/dL (inclusive) (USA sites only: 9.0-10.5, inclusive).
* Stable rhEPO dose for rhEPO users: Group 2 subjects must be using the same rhEPO (epoetins or their biosimilars, or darbepoetin) with total weekly doses that varied by no more than 50% during the 4 weeks prior to Week -4. At Day 1 (randomization), confirm that total weekly doses varied by no more than 50% during the screening period.
* Oral iron therapy: If on oral iron, then doses must not be changed for the 4 weeks prior to Week -4, during the screening phase, and through the first 4 weeks after Randomization.

Exclusion Criteria:

* Dialysis: On dialysis or planning to initiate dialysis during the study.
* Renal transplant: Pre-emptive or scheduled renal transplant.
* High rhEPO dose: An epoetin dose of >=360 IU/kg/week intravenous (IV) or >=250 IU/kg/week subcutaneous (SC) or darbepoetin dose of >=1.8 microgram per kilogram per week (mcg/kg/week) IV or SC within the prior 8 weeks through Day 1 (randomization).
* Use of methoxy polyethylene glycol epoetin beta within the prior 8 weeks through Day 1 (randomization).
* IV iron therapy: Use of IV iron for 4 weeks prior to Screening Week -4, during the screening phase, and through the first 4 weeks after Randomization
* Vitamin B12: Below the lower limit of the reference range (may rescreen in a minimum of 8 weeks).
* Folate: <2.0 nanogram per millilitre (ng/mL) (<4.5 nanomoles per liter [nmol/L]) (may rescreen in a minimum of 4 weeks).
* Ferritin: <40 ng/mL (<40 mcg/L).
* Transferrin saturation (TSAT): Below the lower limit of the reference range
* Myocardial infarction or acute coronary syndrome: Within the 8 weeks prior to Screening through Day 1 (randomization).
* Stroke or transient ischemic attack: Within the 8 weeks prior to Week -4 Screening through Day 1 (randomization).
* Heart failure: Class III/IV heart failure as defined by the New York Heart Association (NYHA) functional classification system diagnosed prior to Week -4 Screening through Day 1 (randomization), symptomatic right heart failure diagnosed prior to Week -4 Screening through Day 1 (randomization).
* Uncontrolled hypertension: Defined as diastolic blood pressure (DBP) >100 mmHg or systolic blood pressure (SBP) >170 mmHg at Week -4 and reconfirmed at Day 1.
* Thrombotic Disease: History of thrombotic disease (e.g., venous thrombosis such as deep vein thrombosis or pulmonary embolism, or arterial thrombosis such as new onset or worsening limb ischemia requiring intervention), except vascular access thrombosis within the 8 weeks prior to Week -4 Screening through Day 1 (randomization).
* Ophthalmology disease: Meeting any ophthalmologic-related exclusion criteria determined at the Screening ophthalmology exam.
* Inflammatory disease: Active chronic inflammatory disease that could impact erythropoiesis (e.g., scleroderma, systemic lupus erythematosis, rheumatoid arthritis, celiac disease) diagnosed prior to Week -4 Screening through Day 1 (randomization).
* Hematological disease: Any hematological disease including those affecting platelets, white or red blood cells (e.g. sickle cell anemia, myelodysplastic syndromes, hematological malignancy, myeloma, hemolytic anemia and thalassemia), coagulation disorders (e.g., antiphospholipid syndrome, Protein C or S deficiency), or any other cause of anemia other than renal disease diagnosed prior to Week -4 Screening through Day 1 (randomization).
* Liver disease: Current liver disease, known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones) or evidence at Screening of abnormal liver function tests [alanine transaminase (ALT) or aspartate transaminase (AST) >2.0 x upper limit of normal (ULN) or total bilirubin >1.5 x ULN]; or other hepatic abnormalities that in the opinion of the investigator would preclude the subject from participation in the study.
* Major surgery: Major surgery (excluding vascular access surgery) within the prior 8 weeks, during the Week -4 Screening phase or planned during the study.
* Transfusion: Blood transfusion within the prior 8 weeks, during the Week -4 Screening phase or an anticipated need for blood transfusion during the study.
* Gastrointestinal (GI) Bleeding: Evidence of actively bleeding peptic, duodenal, or esophageal ulcer disease OR clinically significant GI bleeding within the 8 weeks prior to Week -4 Screening through Day 1 (randomization).
* Acute infection: Clinical evidence of acute infection or history of infection requiring IV antibiotic therapy within the 8 weeks prior to Week -4 Screening through Day 1 (randomization).
* Malignancy: Subjects with a history of malignancy within the prior 5 years, who receiving treatment for cancer, or who have a strong family history of cancer (e.g., familial cancer disorders); with the exception of squamous cell or basal cell carcinoma of the skin that has been definitively treated prior to Week -4 Screening through Day 1 (randomization).
* Severe allergic reactions: History of severe allergic or anaphylactic reactions or hypersensitivity to excipients in the investigational product (see GSK1278863 IB for list of excipients and rhEPO (refer to local product labelling for details).
* Drugs and supplements: Use of any prescription or non-prescription drugs or dietary supplements that are prohibited from Week -4 Screening until the Follow-up Visit.
* Prior investigational product exposure: The Subject has participated in a clinical trial and has received an experimental investigational product within the prior 30 days from Week -4 Screening through Day 1 (randomization).
* Other Conditions: Any other condition, clinical or laboratory abnormality, or examination finding that the Investigator considers would put the subject at unacceptable risk.
* Patient participation: Unwillingness or inability of the subject to follow the procedures or lifestyle or dietary restrictions outlined in the protocol.
* Pregnancy or Lactation: Pregnant females as determined by positive urine human chorionic gonadotropin (hCG) test OR women who are lactating at Week -4 Screening or during the trial.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2013-10-31; Primary Completion 2015-05-01 (Actual); Study Completion 2015-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (111):
- United States (24):
  - GSK Investigational Site, Peoria, Arizona
  - GSK Investigational Site, Azusa, California
  - GSK Investigational Site, La Mesa, California
  - GSK Investigational Site, Laguna Hills, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Dimas, California
  - GSK Investigational Site, West Hills, California
  - GSK Investigational Site, Lauderdale Lakes, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Macon, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Evergreen Park, Illinois
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Farmington, Missouri
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Bethlehem, Pennsylvania
  - GSK Investigational Site, Uniontown, Pennsylvania
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Corsicana, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Temple, Texas
  - GSK Investigational Site, Salt Lake City, Utah
- Australia (4):
  - GSK Investigational Site, Liverpool, New South Wales
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Nedlands, Western Australia
- Canada (8):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Kitchener, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Pointe-Claire, Quebec
- Czechia (7):
  - GSK Investigational Site, Cheb
  - GSK Investigational Site, Liberec
  - GSK Investigational Site, Louny
  - GSK Investigational Site, Mariánské Lázně
  - GSK Investigational Site, Most
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Sokolov
- Denmark (2):
  - GSK Investigational Site, Odense C
  - GSK Investigational Site, Roskilde
- France (7):
  - GSK Investigational Site, Amiens
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Sainte-Foy-lès-Lyon
- Germany (8):
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Demmin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Düsseldorf, North Rhine-Westphalia
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Hungary (2):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Székesfehérvár
- Japan (9):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Gifu
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Shiga
- Poland (5):
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Tarnów
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Zabrze
- Russia (9):
  - GSK Investigational Site, Izhevsk
  - GSK Investigational Site, Kaluga
  - GSK Investigational Site, Khantymansiysk
  - GSK Investigational Site, Krasnodar
  - GSK Investigational Site, Krasnoyarsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Ulyanovsk
  - GSK Investigational Site, Yaroslavl
- South Korea (4):
  - GSK Investigational Site, Anyang-Si Gyeonggi-do
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Daejeon
  - GSK Investigational Site, Gwangju
- Spain (9):
  - GSK Investigational Site, Alcalá de Henares
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, San Sebastián de los Reyes
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Santiago de Compostela
- Sweden (5):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Karlstad
  - GSK Investigational Site, Örebro
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Uppsala
- United Kingdom (8):
  - GSK Investigational Site, Chelmsford
  - GSK Investigational Site, Dorchester
  - GSK Investigational Site, Dundee
  - GSK Investigational Site, Hull
  - GSK Investigational Site, Leeds
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Oxford

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two groups of participants(par.) were enrolled in this study. Group 1 consisted of recombinant human erythropoietin(rhEPO)-naive par. whereas Group 2 consisted of rhEPO users.
Pre-assignment Details: Post screening, eligible par. were randomized to receive either GSK1278863 once a day (QD) or to the Control arm in a 3:1 fashion in Group 1 and 1:1 fashion in Group 2.
Groups:
- rhEPO-Naive GSK1278863: RhEPO-naive participants were randomly assigned to receive GSK1278863 QD for 24 weeks. Participants were blinded to the dose-level they received throughout the study. At Week 24, participants stopped taking GSK1278863, and returned for the follow-up visit at Week 28.
- rhEPO-Naive Control: RhEPO-naive participants were randomly assigned to receive open-label rhEPO (epoetins or their biosimilars, or darbepoetin) as necessary per standard of care, based on the Investigator's clinical judgment, for 24 weeks. At Week 24, participants stopped taking rhEPO (if applicable) and remained off rhEPO or other Erythropoiesis Stimulating Agents (ESA) until at least the follow-up visit at Week 28.
- rhEPO-User GSK1278863: RhEPO users were randomly assigned to receive GSK1278863 QD for 24 weeks. Participants were blinded to the dose-level they received throughout the study. At Week 24, participants stopped taking GSK1278863 and did not re-start rhEPO or other ESAs until after the follow-up visit at Week 28 (except in cases where there was a compelling clinical reason [based on Investigator's opinion] to start rhEPO therapy).
- rhEPO-User Control: RhEPO users were randomly assigned to receive rhEPO (epoetins or their biosimilars, or darbepoetin) as necessary per standard of care, based on the Investigator clinical judgment, for 24 weeks. Participants were allowed to continue rhEPO therapy between Week 24 and 28.
Period: Overall Study
Arm/Group | rhEPO-Naive GSK1278863 | rhEPO-Naive Control | rhEPO-User GSK1278863 | rhEPO-User Control
Started | 136 | 44 | 36 | 36
Completed | 116 | 41 | 32 | 33
Not Completed | 20 | 3 | 4 | 3
Not completed — Adverse Event | 7 | 0 | 2 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 3 | 1 | 0 | 0
Not completed — Reached Defined Stopping Criteria | 2 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 6 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: 252 participants were randomized however the Baseline measurements are provided for the Intent-to-Treat (ITT) population (235 participants), which consisted of all randomized participants who received at least one dose of study drug, had a Baseline and at least one corresponding on-treatment assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | rhEPO-Naive GSK1278863 | rhEPO-Naive Control | rhEPO-User GSK1278863 | rhEPO-User Control | Total
Number analyzed (Participants) | 123 | 43 | 33 | 36 | 235
Age, Continuous [Mean (Standard Deviation); unit: Years] — The Baseline measurement is provided for the Intent-to-Treat (ITT) population, which consisted of all randomized participants who received at least one dose of study drug, had a Baseline and at least one corresponding on-treatment assessment.
  Years | 67.6 (12.21) | 64.3 (14.22) | 62.0 (14.06) | 66.7 (12.89) | 66.1 (13.04)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline measurement is provided for the ITT population.
  Participants
    Female | 75 | 23 | 17 | 23 | 138
    Male | 48 | 20 | 16 | 13 | 97
Race/Ethnicity, Customized [Number; unit: Participants] — Baseline measurement is provided for the ITT population.
  Participants
    African American/African Heritage | 14 | 2 | 2 | 4 | 22
    Central/South Asian Heritage | 0 | 0 | 0 | 1 | 1
    Japanese/East Asian/South East Asian Heritage | 28 | 11 | 9 | 12 | 60
    White | 81 | 30 | 22 | 19 | 152

OUTCOME MEASURES:

1. Primary Outcome: Summary of Hemoglobin (Hgb) Concentration at Week 24
Description: The original Hgb Criteria for Group 1- rhEPO naive participants with a stable baseline Hgb of 8.0-10.0 g/dL (8.0-10.0 g/dL USA site only) and for Group 2- rhEPO users with a stable baseline Hgb of 9.0-10.5 g/dL (9.0-10.5 g/dL USA site only); the Hgb target range was 9.0 to 10.5 g/dL (9.0-10.5 g/dL USA site only). The study amended Hgb Criteria for Group 1- rhEPO naive participants with a stable baseline Hgb of 8.0-11.0 g/dL and Group 2- rhEPO users with a stable baseline Hgb of 9.0-11.5 g/dL; Hgb target range - 10.0 to 11.5 g/dL. Data are presented for those participants following the original criteria ("Original") and those following the amended ("Amended") criteria. The primary objective was to characterize the ability of GSK1278863 to achieve mean Hgb response within the target range.
Time Frame: Week 24
Population: Intent-to-Treat (ITT): The ITT population consisted of all randomized participants who received at least one dose of study drug, had a Baseline and at least one corresponding on-treatment assessment. Only participants who were available at the indicated time point were analyzed.
Measure: Mean (Standard Deviation); unit: grams per deciliter
Arm/Group | rhEPO-Naive GSK1278863 | rhEPO-Naive Control | rhEPO-User GSK1278863 | rhEPO-User Control
Number analyzed (Participants) | 123 | 43 | 33 | 36
grams per deciliter
  Original n=45,15,19,13 | 10.20 (0.906) | 10.64 (0.664) | 10.03 (0.522) | 10.66 (0.620)
  Amended n=61,21,11,17 | 10.96 (1.044) | 11.05 (1.144) | 10.42 (0.827) | 10.86 (1.182)

2. Secondary Outcome: Number of Participants With Hemoglobin (Hgb) in the Target Range at Week 24
Description: Target range is defined as: Original Hgb Criteria of 9.0 to 10.5 gram/deciliter (g/dL), and Amended Hgb Criteria of 10.0 to 11.5 g/dL. Sites in the USA used 9.0 to 10.5 g/dL.
Time Frame: Week 24
Population: ITT population. Only participants who were available at the indicated time point were analyzed.
Measure: Number; unit: participants
Arm/Group | rhEPO-Naive GSK1278863 | rhEPO-Naive Control | rhEPO-User GSK1278863 | rhEPO-User Control
Number analyzed (Participants) | 106 | 36 | 30 | 30
participants | 78 | 20 | 22 | 19

3. Secondary Outcome: Number of Participants Reaching Pre-defined Hgb Stopping Criteria
Description: The Hgb stopping criteria was a value of <7.5 mg/dL obtained on-site via a validated point-of-care Hgb measurement device, which necessitated permanent discontinuation of the study medication. None of the participants met the stopping criteria therefore there is no data to present for this outcome measure.
Time Frame: Over a period of 24 Weeks
Population: ITT population.
Measure: Number; unit: Participants
Arm/Group | rhEPO-Naive GSK1278863 | rhEPO-Naive Control | rhEPO-User GSK1278863 | rhEPO-User Control
Number analyzed (Participants) | 136 | 44 | 36 | 36
Participants | 0 | 0 | 0 | 0

4. Secondary Outcome: Percent Change From Baseline in Hepcidin Concentration at Week 24
Description: Baseline is the last pre-dose hepcidin value. Percent change was calculated as 100 multiplied by (exponential of mean change on log scale minus 1). Change was calculated by subtracting the Baseline value from the Week 24 value.
Time Frame: Baseline and Week 24
Population: Intent-to-Treat (ITT) population consisted all randomized participants who received at least one dose of study drug, had a Baseline and at least one corresponding on-treatment assessment. Only participants with available hepcidin values at Baseline and Week 24 were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: percent change in Hepcidin
Arm/Group | rhEPO-Naive GSK1278863 | rhEPO-Naive Control | rhEPO-User GSK1278863 | rhEPO-User Control
Number analyzed (Participants) | 106 | 35 | 30 | 29
percent change in Hepcidin | -19.27 [-28.10 to -9.36] | 6.67 [-13.62 to 31.72] | -9.87 [-28.59 to 13.76] | -17.12 [-33.22 to 2.86]

5. Secondary Outcome: Maximum Observed Change From Baseline in Serum Erythropoietin (EPO)
Description: Blood samples for control arm were collected pre-dose for EPO measurement. Blood samples for GSK1278863 arms were collected on Day 1 (pre-dose ), Week 4 (6-12 hours post-dose ), Week 4 (7-13, 8-14, 9-15, hours post-dose ), Week 8 (pre -dose ), Week 12 (pre -dose ), Week 16 (pre -dose ), Week 20 (pre -dose , 3 hour post-dose ) Week 24 (pre -dose ), and Week 28 (pre -dose ) for EPO measurement. The maximum observed change from baseline in EPO was recorded for each arm. Baseline value for EPO is the pre-dose value on Day 1. Change from Baseline in EPO was calculated as the individual post-baseline values minus the Baseline value.
Time Frame: Baseline to Week 24
Population: ITT population. Only participants having a Baseline EPO measurement and at least one post-baseline EPO measurement were analyzed.
Measure: Mean (Standard Deviation); unit: International Units per liter
Arm/Group | rhEPO-Naive GSK1278863 | rhEPO-Naive Control | rhEPO-User GSK1278863 | rhEPO-User Control
Number analyzed (Participants) | 123 | 42 | 33 | 36
International Units per liter | 7.27 (12.744) | 27.05 (94.999) | 3.69 (20.554) | 25.85 (38.890)

6. Secondary Outcome: Maximum Observed Percent Change From Baseline in Vascular Endothelial Growth Factor (VEGF)
Description: Blood samples for control arm were collected pre-dose for VEGF measurement. Blood samples for GSK1278863 arms were collected on Day 1 (pre-dose ), Week 4 (6-12 hours post-dose ), Week 4 (7-13, 8-14, 9-15, hours post-dose ), Week 8 (pre -dose ), Week 12 (pre -dose ), Week 16 (pre -dose ), Week 20 (pre -dose , 3 hour post-dose ) Week 24 (pre -dose ), and Week 28 (pre -dose ) for VEGF measurement. The maximum observed change from baseline in VEGF was recorded for each arm . Baseline value for VEGF is the pre-dose value on Day 1. Change from Baseline in VEGF was calculated as the individual post-baseline values minus the Baseline value.
Time Frame: Baseline and up to Week 24
Population: ITT population. Only participants with data available at Baseline and a maximum observed change were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: percent change in VEGF concentration
Arm/Group | rhEPO-Naive GSK1278863 | rhEPO-Naive Control | rhEPO-User GSK1278863 | rhEPO-User Control
Number analyzed (Participants) | 123 | 42 | 33 | 36
percent change in VEGF concentration | 76.36 [59.46 to 95.06] | 26.84 [1.73 to 58.15] | 49.99 [28.28 to 75.39] | 40.85 [19.14 to 66.52]

7. Secondary Outcome: Percentage of Time Within, Below, and Above Hemoglobin (Hgb) Target Range, Between Weeks 12 and 24
Description: The number of days a participant's Hgb was within target range was calculated by estimating (using linear interpolation) the number of days within target range between two scheduled Hgb visits. Percentage of time within range for a participant was calculated by dividing the total number of days that Hgb was within range during Weeks 12 to 24 by the total number of days the participant remained on treatment during Weeks 12 to 24. Similary, percent of time above and below Hgb target range was calculated. Target range was defined as: Original Hgb Criteria of 9.0 to 10.5 g/dL, and Amended Hgb Criteria of 10.0 to 11.5 g/dL. Sites in the USA used 9.0 to 10.5 g/dL.
Time Frame: Weeks 12 to 24
Population: ITT population. Only participants with data available at specific time points were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | rhEPO-Naive GSK1278863 | rhEPO-Naive Control | rhEPO-User GSK1278863 | rhEPO-User Control
Number analyzed (Participants) | 112 | 38 | 30 | 32
percentage of days
  Percentage of time within target range | 68.99 (34.612) | 51.01 (41.403) | 75.06 (32.485) | 61.29 (43.352)
  Percentage of time above target range | 22.84 (33.825) | 45.10 (42.579) | 17.96 (28.809) | 31.10 (41.683)
  Percentage of time below target range | 8.17 (20.301) | 3.89 (16.175) | 6.98 (21.118) | 7.61 (25.113)

8. Secondary Outcome: Change From Baseline in Ferritin Concentration at Week 24
Description: Baseline is the last pre-dose ferritin value. Change was calculated by subtracting the Baseline value from the Week 24 value.
Time Frame: Baseline and Week 24
Population: ITT population. Only participants with data available at specific time point were analyzed.
Measure: Mean (Standard Deviation); unit: micrograms per liter
Arm/Group | rhEPO-Naive GSK1278863 | rhEPO-Naive Control | rhEPO-User GSK1278863 | rhEPO-User Control
Number analyzed (Participants) | 108 | 36 | 30 | 30
micrograms per liter | -30.8 (110.50) | -2.4 (77.06) | -63.4 (141.93) | -20.4 (63.38)

9. Secondary Outcome: Change From Baseline in Transferrin Concentration at Week 24
Description: Baseline is the last pre-dose transferrin value. Change from Baseline in transferrin was calculated by subtracting the Baseline value from the Week 24 value.
Time Frame: Baseline and Week 24
Population: ITT population. Only participants with data available at specific time point were analyzed.
Measure: Mean (Standard Deviation); unit: grams per liter
Arm/Group | rhEPO-Naive GSK1278863 | rhEPO-Naive Control | rhEPO-User GSK1278863 | rhEPO-User Control
Number analyzed (Participants) | 107 | 36 | 30 | 30
grams per liter | 0.077 (0.3577) | -0.008 (0.2694) | 0.171 (0.4124) | 0.018 (0.2395)

10. Secondary Outcome: Percent Change From Baseline in Transferrin Saturation at Week 24
Description: Transferrin saturation is measured as a percentage; it is a ratio of serum iron and total iron-binding capacity. Baseline is the last pre-dose transferrin saturation value. Percent change was calculated as 100 multiplied by (exponential of mean change on log scale minus 1). Change was calculated by subtracting the Baseline value from the post-dose value.
Time Frame: Baseline and Week 24
Population: ITT population. Only participants with data available at specific time point were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Arm/Group | rhEPO-Naive GSK1278863 | rhEPO-Naive Control | rhEPO-User GSK1278863 | rhEPO-User Control
Number analyzed (Participants) | 106 | 35 | 30 | 30
percent change | -1.1 [-8.0 to 6.4] | 12.3 [2.2 to 23.3] | -15.7 [-26.8 to -3.0] | 11.4 [-14.7 to 45.6]

11. Secondary Outcome: Change From Baseline in Total Iron at Week 24
Description: Baseline is the last pre-dose total iron value. Change from Baseline was calculated by subtracting the Baseline value from the Week 24 value.
Time Frame: Baseline and Week 24
Population: ITT population. Only participants with available total iron values at Baseline and Week 24 were analyzed.
Measure: Mean (Standard Deviation); unit: micromoles per liter
Arm/Group | rhEPO-Naive GSK1278863 | rhEPO-Naive Control | rhEPO-User GSK1278863 | rhEPO-User Control
Number analyzed (Participants) | 107 | 36 | 30 | 30
micromoles per liter | 1.0 (5.01) | 2.5 (5.98) | -1.8 (5.54) | 0.7 (8.36)

12. Secondary Outcome: Change From Baseline in Total Iron Binding Capacity (TIBC) at Week 24
Description: TIBC measures the blood's capacity to bind iron with transferrin. Baseline is the last pre-dose TIBC value. Change from Baseline in TIBC was calculated by subtracting the Baseline value from the Week 24 value.
Time Frame: Baseline and Week 24
Population: ITT population. Only participants with data available at specific timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: micromoles per liter
Arm/Group | rhEPO-Naive GSK1278863 | rhEPO-Naive Control | rhEPO-User GSK1278863 | rhEPO-User Control
Number analyzed (Participants) | 106 | 35 | 30 | 30
micromoles per liter | 3.2 (6.46) | 0.1 (5.17) | 3.0 (9.44) | -1.0 (6.69)

13. Secondary Outcome: Change From Baseline in Reticulocyte Hemoglobin (CHr) at Week 24
Description: Reticulocytes are slightly immature red blood cells. Reticulocyte Hgb content is used to differentiate iron deficiency from other causes of anemia. Baseline is the last pre-dose CHr value. Change from Baseline in reticulocyte Hgb was calculated by subtracting the Baseline value from the post-dose value.
Time Frame: Baseline and Week 24
Population: ITT population. Only participants with data available at specific time point were analyzed.
Measure: Mean (Standard Deviation); unit: picogram
Arm/Group | rhEPO-Naive GSK1278863 | rhEPO-Naive Control | rhEPO-User GSK1278863 | rhEPO-User Control
Number analyzed (Participants) | 108 | 35 | 30 | 30
picogram | -0.19 (1.109) | -0.33 (1.085) | -0.32 (0.864) | -0.19 (1.546)

14. Secondary Outcome: Change From Baseline in Hematocrit at Week 24
Description: Baseline is the last pre-dose hematocrit value. Change from Baseline was calculated by subtracting the Baseline value from the Week 24 value.
Time Frame: Baseline and Week 24
Population: ITT population. Only participants with data available at specific timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change in Fraction of 1
Arm/Group | rhEPO-Naive GSK1278863 | rhEPO-Naive Control | rhEPO-User GSK1278863 | rhEPO-User Control
Number analyzed (Participants) | 111 | 36 | 30 | 30
percentage change in Fraction of 1 | 2.64 (3.389) | 3.13 (3.245) | -0.66 (3.074) | 2.09 (3.243)

15. Secondary Outcome: Change From Baseline in Red Blood Cell Count at Week 24
Description: Baseline is the last pre-dose red blood cell count. Change from Baseline in red blood cell count was calculated by subtracting the Baseline count from the post-dose count.
Time Frame: Baseline and Week 24
Population: ITT population. Only participants with data available at specific time point were analyzed.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | rhEPO-Naive GSK1278863 | rhEPO-Naive Control | rhEPO-User GSK1278863 | rhEPO-User Control
Number analyzed (Participants) | 111 | 36 | 30 | 30
10^12 cells per liter | 0.28 (0.377) | 0.34 (0.365) | -0.08 (0.312) | 0.22 (0.318)

16. Secondary Outcome: Change From Baseline in Reticulocyte Cell Count at Week 24
Description: Reticulocyte count is a blood test that measures the percentage of reticulocytes in the blood. Reticulocytes are slightly immature red blood cells. Baseline is the last pre-dose red reticulocyte count. Change from Baseline in reticulocyte cell count was calculated by subtracting the Baseline count from the Week 24 count.
Time Frame: Baseline and Week 24
Population: ITT population. Only participants with data available at specific timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of reticulocytes
Arm/Group | rhEPO-Naive GSK1278863 | rhEPO-Naive Control | rhEPO-User GSK1278863 | rhEPO-User Control
Number analyzed (Participants) | 111 | 36 | 30 | 31
percentage of reticulocytes | -0.02 (0.551) | -0.12 (0.648) | 0.27 (0.892) | -0.09 (0.755)

17. Secondary Outcome: Concentration of GSK1278863 and Relevant Metabolites as a Population Pharmacokinetic Endpoint
Description: Blood samples were collected for individual plasma GSK1278863 and metabolite (GSK2391220, GSK2487818, GSK2506102, GSK2531398, GSK2531401, and GSK2531403) concentration measurement on Day 1 (pre-dose), Wk 4 (6-12 hour, 7-13 hour, 8-14 hour, 9-15 hour post-dose), and Wk 20 (pre-dose, 1 hour, 2 hour, 3 hour post-dose). Participants available in each arm at the specified time points have been presented.
Time Frame: Day 1 (pre-dose), Week (Wk) 4 (6-12 hour, 7-13 hour, 8-14 hour, 9-15 hour post-dose), and Wk 20 (pre-dose, 1 hour, 2 hour, 3 hour post-dose)
Population: Pharmacokinetics (PK) population: All participants from whom a PK sample was obtained and analyzed. This population did not include participants from the control groups.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | rhEPO-Naive GSK1278863 | rhEPO-User GSK1278863
Number analyzed (Participants) | 134 | 35
nanograms per milliliter
  GSK1278863, Day 1, Pre-Dose, n=128, 35 | 0.0 (0.00) | 0.0 (0.00)
  GSK1278863, Wk 4, 6-12 hour Post-Dose, n=116, 31 | 2.0 (5.18) | 1.1 (1.69)
  GSK1278863, Wk 4, 7-13 hour Post-Dose, n=117, 31 | 2.3 (7.06) | 0.8 (1.22)
  GSK1278863, Wk 4, 8-14 hour Post-Dose, n=116, 31 | 1.6 (4.93) | 1.6 (5.49)
  GSK1278863, Wk 4, 9-15 hour Post-Dose, n=116, 31 | 1.4 (4.52) | 1.6 (4.60)
  GSK1278863, Wk 20, Pre-Dose, n=111, 29 | 0.6 (3.07) | 0.3 (0.92)
  GSK1278863, Wk 20, 1 hour Post-Dose, n=110, 28 | 22.8 (35.93) | 19.8 (19.66)
  GSK1278863, Wk 20, 2 hour Post-Dose, n=109, 29 | 17.0 (28.57) | 19.4 (21.92)
  GSK1278863, Wk 20, 3 hour Post-Dose, n=109, 29 | 11.6 (19.56) | 13.9 (19.12)
  GSK2391220, Day 1, Pre-Dose, n=128, 35 | 0.0 (0.00) | 0.0 (0.00)
  GSK2391220, Wk 4, 6-12 hour Post-Dose, n=116, 31 | 3.2 (5.21) | 3.7 (2.89)
  GSK2391220, Wk 4, 7-13 hour Post-Dose, n=117, 31 | 3.1 (5.67) | 3.2 (2.43)
  GSK2391220, Wk 4, 8-14 hour Post-Dose, n=116, 31 | 2.8 (5.01) | 2.9 (2.54)
  GSK2391220, Wk 4, 9-15 hour Post-Dose, n=116, 31 | 2.6 (4.89) | 3.1 (2.76)
  GSK2391220, Wk 20, Pre-Dose, n=111, 29 | 1.0 (2.06) | 0.8 (0.98)
  GSK2391220, Wk 20, 1 hour Post-Dose, n=110, 28 | 2.1 (3.52) | 1.6 (1.39)
  GSK2391220, Wk 20, 2 hour Post-Dose, n=109, 29 | 3.8 (5.08) | 3.7 (2.98)
  GSK2391220, Wk 20, 3 hour Post-Dose, n=109, 29 | 4.5 (5.43) | 4.7 (3.53)
  GSK2487818, Day 1, Pre-Dose, n=128, 35 | 0.0 (0.00) | 0.0 (0.00)
  GSK2487818, Wk 4, 6-12 hour Post-Dose, n=116, 31 | 1.2 (3.87) | 1.0 (0.96)
  GSK2487818, Wk 4, 7-13 hour Post-Dose, n=116, 31 | 1.1 (4.11) | 0.7 (0.70)
  GSK2487818, Wk 4, 8-14 hour Post-Dose, n=116, 31 | 1.0 (4.48) | 0.6 (0.66)
  GSK2487818, Wk 4, 9-15 hour Post-Dose, n=116, 31 | 0.9 (4.09) | 0.8 (1.16)
  GSK2487818, Wk 20, Pre-Dose, n=111, 29 | 0.2 (0.56) | 0.1 (0.31)
  GSK2487818, Wk 20, 1 hour Post-Dose, n=110, 28 | 1.4 (3.07) | 1.0 (1.09)
  GSK2487818, Wk 20, 2 hour Post-Dose, n=109, 29 | 2.8 (4.28) | 2.7 (2.21)
  GSK2487818, Wk 20, 3 hour Post-Dose, n=109, 29 | 3.1 (4.07) | 3.1 (2.56)
  GSK2506102, Day 1, Pre-Dose, n=128, 35 | 0.0 (0.00) | 0.0 (0.00)
  GSK2506102, Wk 4, 6-12 hour Post-Dose, n=116, 31 | 1.0 (1.30) | 1.2 (0.65)
  GSK2506102, Wk 4, 7-13 hour Post-Dose, n=117, 31 | 1.0 (1.51) | 1.1 (0.61)
  GSK2506102, Wk 4, 8-14 hour Post-Dose, n=116, 31 | 0.9 (1.19) | 1.0 (0.61)
  GSK2506102, Wk 4, 9-15 hour Post-Dose, n=116, 31 | 0.9 (1.29) | 1.1 (0.69)
  GSK2506102, Wk 20, Pre-Dose, n=111, 29 | 0.4 (0.73) | 0.4 (0.42)
  GSK2506102, Wk 20, 1 hour Post-Dose, n=110, 28 | 0.6 (0.88) | 0.5 (0.40)
  GSK2506102, Wk 20, 2 hour Post-Dose, n=109, 29 | 0.9 (1.15) | 1.0 (0.71)
  GSK2506102, Wk 20, 3 hour Post-Dose, n=109, 29 | 1.1 (1.25) | 1.2 (0.88)
  GSK2531398, Day 1, Pre-Dose, n=128, 35 | 0.0 (0.01) | 0.0 (0.00)
  GSK2531398, Wk 4, 6-12 hour Post-Dose, n=116, 31 | 1.3 (2.06) | 1.4 (1.08)
  GSK2531398, Wk 4, 7-13 hour Post-Dose, n=117, 31 | 1.2 (2.50) | 1.2 (0.99)
  GSK2531398, Wk 4, 8-14 hour Post-Dose, n=116, 31 | 1.1 (2.01) | 1.1 (0.93)
  GSK2531398, Wk 4, 9-15 hour Post-Dose, n=116, 31 | 1.0 (2.10) | 1.2 (1.12)
  GSK2531398, Wk 20, Pre-Dose, n=111, 29 | 0.3 (0.87) | 0.3 (0.38)
  GSK2531398, Wk 20, 1 hour Post-Dose, n=110, 28 | 0.8 (1.53) | 0.6 (0.54)
  GSK2531398, Wk 20, 2 hour Post-Dose, n=109, 29 | 1.6 (2.31) | 1.5 (1.22)
  GSK2531398, Wk 20, 3 hour Post-Dose, n=109, 29 | 2.0 (2.42) | 2.0 (1.57)
  GSK2531401, Day 1, Pre-Dose, n=128, 35 | 0.0 (0.00) | 0.0 (0.00)
  GSK2531401, Wk 4, 6-12 hour Post-Dose, n=116, 31 | 2.8 (4.00) | 4.3 (2.55)
  GSK2531401, Wk 4, 7-13 hour Post-Dose, n=117, 31 | 2.7 (3.58) | 4.0 (2.29)
  GSK2531401, Wk 4, 8-14 hour Post-Dose, n=116, 31 | 2.7 (3.74) | 3.8 (2.31)
  GSK2531401, Wk 4, 9-15 hour Post-Dose, n=116, 31 | 2.5 (3.53) | 3.8 (2.29)
  GSK2531401, Wk 20, Pre-Dose, n=111, 29 | 1.3 (2.41) | 1.4 (1.38)
  GSK2531401, Wk 20, 1 hour Post-Dose, n=110, 28 | 1.6 (2.65) | 1.6 (1.29)
  GSK2531401, Wk 20, 2 hour Post-Dose, n=109, 29 | 2.3 (3.14) | 2.5 (1.85)
  GSK2531401, Wk 20, 3 hour Post-Dose, n=109, 29 | 2.8 (3.50) | 3.2 (2.22)
  GSK2531403, Day 1, Pre-Dose, n=128, 35 | 0.0 (0.00) | 0.0 (0.00)
  GSK2531403, Wk 4, 6-12 hour Post-Dose, n=116, 31 | 3.7 (5.43) | 4.5 (3.14)
  GSK2531403, Wk 4, 7-13 hour Post-Dose, n=117, 31 | 3.5 (5.27) | 3.9 (2.56)
  GSK2531403, Wk 4, 8-14 hour Post-Dose, n=116, 31 | 3.4 (5.68) | 3.7 (2.72)
  GSK2531403, Wk 4, 9-15 hour Post-Dose, n=116, 31 | 3.2 (5.42) | 3.8 (3.01)
  GSK2531403, Wk 20, Pre-Dose, n=111, 29 | 1.4 (2.65) | 1.2 (1.25)
  GSK2531403, Wk 20, 1 hour Post-Dose, n=110, 28 | 2.3 (3.69) | 1.9 (1.38)
  GSK2531403, Wk 20, 2 hour Post-Dose, n=109, 29 | 3.9 (5.03) | 3.8 (2.95)
  GSK2531403, Wk 20, 3 hour Post-Dose, n=109, 29 | 4.7 (5.43) | 4.9 (3.75)

18. Secondary Outcome: Mean Number of Dose Adjustments up to 24 Weeks
Description: After 4 Weeks, the need to adjust the dose of GSK1278863 was evaluated at every scheduled visit, to maintain hemoglobin within the target range. Target range was defined as: Original Hgb Criteria of 9.0 to 10.5 g/dL, and Amended Hgb Criteria of 10.0 to 11.5 g/dL. Sites in the USA used 9.0 to 10.5 g/dL. Dose adjustments were assigned automatically via the interactive voice/web response system.
Time Frame: From Week 4 up to 24 Weeks
Population: Intent-to-Treat population. Only those participants with at least one dose adjustment of GSK1278863 were analyzed.
Measure: Mean (Standard Deviation); unit: number of adjustments
Arm/Group | rhEPO-Naive GSK1278863 | rhEPO-User GSK1278863
Number analyzed (Participants) | 102 | 26
number of adjustments | 1.8 (0.82) | 1.7 (0.72)

19. Secondary Outcome: Number of Participants With Dose Adjustments up to 24 Weeks, as a Measure of Dose Adjustment Frequency
Description: After 4 Weeks, the need to adjust the dose of GSK1278863 was evaluated at every scheduled visit, to maintain hemoglobin within the target range. Target range was defined as: Original Hgb Criteria of 9.0 to 10.5 g/dL, and Amended Hgb Criteria of 10.0 to 11.5 g/dL. Sites in the USA used 9.0 to 10.5 g/dL. Dose adjustments were assigned automatically via the interactive voice/web response system. Frequency is presented as the number of participants with dose adjustment(s) once, twice, thrice, four times, or five times.
Time Frame: From week 4 up to 24 weeks
Population: Intent-to-Treat population. Only those participants with at least one dose adjustment of GSK1278863 were analyzed.
Measure: Number; unit: participants
Arm/Group | rhEPO-Naive GSK1278863 | rhEPO-User GSK1278863
Number analyzed (Participants) | 102 | 26
participants
  Once | 39 | 11
  Twice | 50 | 11
  Thrice | 8 | 4
  Four times | 4 | 0
  Five times or more | 1 | 0

20. Secondary Outcome: Timing of Dose Adjustments at Weeks 4, 8, 12, 16, and 20
Description: After 4 Weeks, the need to adjust the dose of GSK1278863 was evaluated at every scheduled visit, to maintain hemoglobin within the target range. Target range was defined as: Original Hgb Criteria of 9.0 to 10.5 g/dL, and Amended Hgb Criteria of 10.0 to 11.5 g/dL. Sites in the USA used 9.0 to 10.5 g/dL. Dose adjustments were assigned automatically via the interactive voice/web response system. The number of participants with an adjustment are presented at the timings at which adjustments were done.
Time Frame: From Week 4 up to Week 20
Population: ITT population. Only those participants with at least one dose adjustment of GSK1278863 were analyzed.
Measure: Number; unit: Participants
Arm/Group | rhEPO-Naive GSK1278863 | rhEPO-User GSK1278863
Number analyzed (Participants) | 102 | 26
Participants
  Week 4 | 78 | 21
  Week 8 | 24 | 6
  Week 12 | 30 | 7
  Week 16 | 30 | 6
  Week 20 | 22 | 5

21. Secondary Outcome: Mean Total Cumulative Dose of GSK1278863 up to 24 Weeks
Description: The starting dose was kept constant for the first 4 Weeks after randomization. Later, the need to adjust the dose of GSK1288863 was evaluated at every scheduled visit according to a pre-specified algorithm, to achieve and maintain hemoglobin within the specified target range. Target range was defined as: Original Hgb Criteria of 9.0 to 10.5 g/dL, and Amended Hgb Criteria of 10.0 to 11.5 g/dL. Sites in the USA used 9.0 to 10.5 g/dL.
Time Frame: Up to 24 Weeks
Population: ITT population.
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | rhEPO-Naive GSK1278863 | rhEPO-User GSK1278863
Number analyzed (Participants) | 123 | 33
milligrams | 249.75 (186.921) | 320.42 (214.865)

22. Secondary Outcome: Mean Final Dose of GSK1278863 up to 24 Weeks
Description: as for outcome 21
Time Frame: Up to 24 Weeks
Population: ITT population.
Measure: Mean (Standard Deviation); unit: milligrams per day
Arm/Group | rhEPO-Naive GSK1278863 | rhEPO-User GSK1278863
Number analyzed (Participants) | 123 | 33
milligrams per day | 1.75 (1.809) | 1.86 (1.692)

23. Secondary Outcome: Number of Hemoglobin (Hgb) Excursions
Description: A Hgb excursion is a series of decreasing or increasing Hgb values differing by >=1.5 grams per deciliter. Hgb cycle is calculated as two consecutive Hgb excursions in different directions.
Time Frame: Up to 24 Weeks.
Population: Completers Population: ITT participants who fully completed study without prematurely discontinuing study drug. Only participants with Hgb excursions were analyzed.
Measure: Number; unit: number of excursions
Arm/Group | rhEPO-Naive GSK1278863 | rhEPO-Naive Control | rhEPO-User GSK1278863 | rhEPO-User Control
Number analyzed (Participants) | 23 | 10 | 4 | 8
number of excursions | 26 | 10 | 4 | 9

24. Secondary Outcome: Number of Hemoglobin (Hgb) Cycles up to 24 Weeks
Description: A Hgb cycle is calculated as two consecutive Hgb excursions in different directions. A Hgb excursion is a series of decreasing or increasing Hgb values differing by >=1.5 grams per deciliter.
Time Frame: Up to 24 Weeks
Population: Completers population. Only participants with Hgb cycles were analyzed.
Measure: Number; unit: number of Hgb cycles
Arm/Group | rhEPO-Naive GSK1278863 | rhEPO-Naive Control | rhEPO-User GSK1278863 | rhEPO-User Control
Number analyzed (Participants) | 3 | 0 | 0 | 0
number of Hgb cycles | 3 |  |  |

25. Secondary Outcome: Number of Dose Cycles up to 24 Weeks
Description: A dose cycle is a series of three directional dose changes (that is, increase, decrease, increase; or decrease, increase, decrease).
Time Frame: Up to 24 weeks
Population: Completers population. Only participants in the GSK1278863 arms with dose cycles were analyzed.
Measure: Number; unit: number
Arm/Group | rhEPO-Naive GSK1278863 | rhEPO-User GSK1278863
Number analyzed (Participants) | 1 | 0
number | 1 |

26. Secondary Outcome: Number of Participants With at Least One Hemoglobin (Hgb) Excursion up to 24 Weeks.
Description: A Hgb excursion is a series of decreasing or increasing Hgb values differing by >=1.5 grams per deciliter.
Time Frame: Up to 24 weeks
Population: Completers population.
Measure: Number; unit: participants
Arm/Group | rhEPO-Naive GSK1278863 | rhEPO-Naive Control | rhEPO-User GSK1278863 | rhEPO-User Control
Number analyzed (Participants) | 106 | 36 | 30 | 30
participants | 23 | 10 | 4 | 8

27. Secondary Outcome: Number of Participants With at Least One Hemoglobin (Hgb) Cycle up to 24 Weeks
Description: A Hgb excursion is a series of decreasing or increasing Hgb values differing by >=1.5 grams per deciliter. A Hgb cycle is two consecutive Hgb excursions in different directions.
Time Frame: Up to 24 weeks
Population: Completers population.
Measure: Number; unit: participants
Arm/Group | rhEPO-Naive GSK1278863 | rhEPO-Naive Control | rhEPO-User GSK1278863 | rhEPO-User Control
Number analyzed (Participants) | 106 | 36 | 30 | 30
participants | 3 | 0 | 0 | 0

28. Secondary Outcome: Number of Participants With at Least One Dose Cycle up to 24 Weeks
Description: A dose cycle is a series of three directional dose changes (that is, increase, decrease, increase; or decrease, increase, decrease). participants
Time Frame: Up to 24 weeks
Population: Completers population. Only participants in the GSK1278863 arms with dose cycles were analyzed.
Measure: Number; unit: participants
Arm/Group | rhEPO-Naive GSK1278863 | rhEPO-User GSK1278863
Number analyzed (Participants) | 106 | 30
participants | 1 | 0

29. Secondary Outcome: Number of Participants Receiving Additional Therapies of Blood Transfusions, Intravenous (IV) Iron or rhEPO at Any Time Post-Baseline
Description: Participants receiving additional therapies of blood transfusions, intravenous (IV) iron or rhEPO any time Post Baseline were analyzed. RhEPO was not applicable for the control arms since it was a planned therapy in those arms, hence presented as NA. (EudraCT only: A value of 99999 is used where no data is available or NA.)
Time Frame: From Day 1 up to Week 28
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | rhEPO-Naive GSK1278863 | rhEPO-Naive Control | rhEPO-User GSK1278863 | rhEPO-User Control
Number analyzed (Participants) | 123 | 43 | 33 | 36
participants
  Blood Transfusions | 3 | 1 | 1 | 0
  IV Iron | 20 | 3 | 3 | 4
  Inadvertent rhEPO use | 4 | NA — Non-rhEPO users were not evaluated for this data point. | 9 | NA — Non-rhEPO users were not evaluated for this data point.
  Rescue rhEPO | 1 | NA — Non-rhEPO users were not evaluated for this data point. | 0 | NA — Non-rhEPO users were not evaluated for this data point.

30. Secondary Outcome: Number of Weeks Dose Withheld Because Hemoglobin (Hgb) Exceeded the Upper Limit
Description: Number of Weeks dose was withheld because hemoglobin exceed the upper limit is presented as the number of participants with withheld dose during the time periods categorized by Weeks.
Time Frame: From Week 4 up to Week 24
Population: ITT population.
Measure: Number; unit: participants
Arm/Group | rhEPO-Naive GSK1278863 | rhEPO-User GSK1278863
Number analyzed (Participants) | 123 | 33
participants
  0 Weeks | 102 | 30
  >0-4 Weeks | 4 | 2
  >4-8 Weeks | 8 | 0
  >8-12 Weeks | 8 | 0
  >12 Weeks | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAEs) were collected from the start of study treatment until the follow-up contact (up to 28 weeks).
Description: AEs and SAEs were collected from participants of the safety population, comprised of all participants who received at least one dose of study drug.
Arm/Group | rhEPO-Naive GSK1278863 | rhEPO-Naive Control | rhEPO-User GSK1278863 | rhEPO-User Control
Serious Adverse Events (participants affected / at risk) | 23/134 | 7/45 | 7/36 | 7/35
Other Adverse Events (participants affected / at risk) | 47/134 | 14/45 | 20/36 | 13/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | rhEPO-Naive GSK1278863 (N=134) | rhEPO-Naive Control (N=45) | rhEPO-User GSK1278863 (N=36) | rhEPO-User Control (N=35)
ANY EVENT (Renal and urinary disorders) | 2 | 3 | 2 | 3
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 2 | 2 | 1 | 1
GLOMERULONEPHRITIS CHRONIC (Renal and urinary disorders) | 0 | 0 | 1 | 0
DIABETIC NEPHROPATHY (Renal and urinary disorders) | 0 | 1 | 0 | 0
RENAL FAILURE (Renal and urinary disorders) | 0 | 0 | 0 | 1
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 | 0 | 0 | 1
ANY EVENT (Infections and infestations) | 2 | 3 | 1 | 1
PNEUMONIA (Infections and infestations) | 1 | 1 | 1 | 0
PYELONEPHRITIS CHRONIC (Infections and infestations) | 1 | 0 | 0 | 0
APPENDICITIS (Infections and infestations) | 0 | 1 | 0 | 0
CELLULITIS (Infections and infestations) | 0 | 1 | 0 | 0
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 0 | 0 | 0 | 1
ANY EVENT (Cardiac disorders) | 4 | 1 | 0 | 1
ANGINA PECTORIS (Cardiac disorders) | 1 | 0 | 0 | 0
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 1 | 0 | 0 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 | 0 | 0 | 1
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 | 0 | 0 | 0
CARDIAC FAILURE (Cardiac disorders) | 0 | 1 | 0 | 0
ANY EVENT (Gastrointestinal disorders) | 1 | 0 | 1 | 1
GASTRIC ULCER (Gastrointestinal disorders) | 1 | 0 | 0 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 0 | 1 | 0
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 1
ANY EVENT (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0
FLUID OVERLOAD (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
ANY EVENT (Nervous system disorders) | 1 | 0 | 1 | 1
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 1 | 0 | 0 | 0
CEREBRAL MICROANGIOPATHY (Nervous system disorders) | 0 | 0 | 1 | 0
NEURALGIA (Nervous system disorders) | 0 | 0 | 0 | 1
ANY EVENT (Vascular disorders) | 2 | 0 | 1 | 0
DIABETIC VASCULAR DISORDER (Vascular disorders) | 0 | 0 | 1 | 0
HYPERTENSION (Vascular disorders) | 1 | 0 | 0 | 0
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1 | 0 | 0 | 0
ANY EVENT (Investigations) | 2 | 0 | 0 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0 | 0
FALSE POSITIVE INVESTIGATION RESULT (Investigations) | 1 | 0 | 0 | 0
ANY EVENT (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
CHONDROCALCINOSIS PYROPHOSPHATE (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
ANY EVENT (Psychiatric disorders) | 2 | 0 | 0 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 1 | 0 | 0 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 | 0 | 0 | 0
ANY EVENT (General disorders) | 0 | 0 | 0 | 1
CHEST PAIN (General disorders) | 0 | 0 | 0 | 1
ANY EVENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
HEPATIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
ANY EVENT (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0
Biliary sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0
Shunt malfunction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | rhEPO-Naive GSK1278863 (N=134) | rhEPO-Naive Control (N=45) | rhEPO-User GSK1278863 (N=36) | rhEPO-User Control (N=35)
NASOPHARYNGITIS (Infections and infestations) | 15 | 2 | 7 | 2
CONJUNCTIVITIS (Infections and infestations) | 1 | 0 | 2 | 0
BRONCHITIS (Infections and infestations) | 2 | 1 | 0 | 3
DIARRHOEA (Gastrointestinal disorders) | 10 | 0 | 0 | 6
NAUSEA (Gastrointestinal disorders) | 8 | 1 | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 5 | 1 | 1 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 3
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 2
OEDEMA PERIPHERAL (General disorders) | 5 | 0 | 2 | 3
FATIGUE (General disorders) | 3 | 1 | 1 | 2
HYPERKALAEMIA (Metabolism and nutrition disorders) | 2 | 0 | 2 | 1
GOUT (Metabolism and nutrition disorders) | 2 | 0 | 1 | 2
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 4 | 0 | 0
HYPERTENSION (Vascular disorders) | 2 | 1 | 4 | 1
BLOOD PRESSURE INCREASED (Investigations) | 1 | 0 | 1 | 2
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 2
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 3 | 0
Asthenia (General disorders) | 1 | 3 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.